CLINICAL TRIAL: NCT04430036
Title: A Phase II Trial of Neoadjuvant AGEN1884 Plus AGEN2034 in Combination With Cisplatin-Gemcitabine for Muscle-Invasive Bladder Cancer Prior to Radical Cystectomy
Brief Title: AGEN1884 Plus AGEN2034 Combined With Cisplatin-Gemcitabine for Muscle-Invasive Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 19-0193; HSC20200027H (Other: UT Health Science Center San Antonio IRB)
Record Dates: First submitted 2020-05-08; First posted 2020-06-12 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Urinary Bladder Neoplasms
Keywords: muscle-invasive, non-metastatic
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — balstilimab; spartalizumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: This is a phase II trial to evaluate the tolerability, efficacy, and immune outcomes of AGEN1884 plus AGEN2034 concurrent with cisplatin and gemcitabine in the neoadjuvant treatment of muscle-invasive, non-metastatic bladder cancer prior to radical cystectomy. We will begin with an initial safety run-in to establish the safety of the combination prior to expansion to the full planned phase II. The overall phase II will be an open-label, single arm study in two stages to evaluate the efficacy of the combination in pathologic downstaging of MIBC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cisplatin, Gemcitabine plus human monoclonal antibodies (Experimental): The safety run-in of the study will first enroll three patients who will begin treatment with cisplatin and gemcitabine plus AGEN2034 and AGEN1884 as outlined in the treatment plan. These first 3 patients will be assessed for DLTs and there will be a pause in enrollment until all three complete the DLT period. If there are no DLTs in the first 3 patients, we will proceed to further accrual to stage I of phase II. If there is 1 DLT in the initial 3 patients, we will enroll 3 additional patients to the safety run-in. If > 2 DLTs are experienced in the initial 3 patients, the study will be terminated, otherwise additional subjects will be enrolled into the phase ll first stage and reassessed after 2 cycles of therapy and proceed to planned surgery. If criteria are met to continue to the second stage of the Phase II portion of the study, additional patients will be enrolled for an anticipated total of 36 evaluable patients. Patients will be treated and endpoints evaluated.
  Interventions: Drug: AGEN1884; Drug: AGEN2034; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: AGEN1884 — A fully human monoclonal Anti-PD-1 Antibody
  Other Names: anti-CTLA-4 antibody
Drug: AGEN2034 — A fully human monoclonal Anti-PD-1 Antibody
  Other Names: Anti-PD-1
Drug: Cisplatin — Alkylating antineoplastic agent
  Other Names: Gemzar, Platinol® and Platinol®-AQ
Drug: Gemcitabine — Antimetabolite antineoplastic agent
  Other Names: Gebina, Gemalata, Gembin, Gembine, Gembio, Gemcel, Gemcetin

SUMMARY:
This is a phase II trial to evaluate the tolerability, efficacy, and immune outcomes of AGEN1884 plus AGEN2034 concurrent with cisplatin and gemcitabine in the neoadjuvant treatment of muscle-invasive, non-metastatic bladder cancer prior to radical cystectomy.

DETAILED DESCRIPTION:
We will begin with an initial safety run-in to establish the safety of the combination prior to expansion to the full planned phase II. The overall phase II will be an open-label, single arm study in two stages to evaluate the efficacy of the combination in pathologic downstaging of MIBC. Patients will receive four 21-day cycles of neoadjuvant therapy consisting of cisplatin and gemcitabine plus AGEN2034 in all 4 cycles and AGEN1884 in cycles 1 and 3. Patients will proceed to radical cystectomy within 10 weeks after the final dose of this therapy. The primary endpoint of pathologic tumor downstaging will be assessed at the time of cystectomy.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of muscle-invasive, non-metastatic urothelial carcinoma of the bladder, cT2-4, N0-1, M0
2. Eligible to receive cisplatin-based chemotherapy, with eligibility defined as meeting all of the following criteria:

   1. Eastern Cooperative Oncology Group performance status of ¬0-1
   2. Creatinine clearance (CrCl) of >50 mL/min, as measured by 24-hour urine collection or estimated by the CKD-EPI equation. Patients with CrCl between 50 - 60 mL/min are eligible for the study but will receive split dose cisplatin
   3. Grade < 2 hearing loss
   4. Grade < 2 peripheral neuropathy
   5. New York Heart Association Class < III heart failure
3. Eligible to receive gemcitabine as dosed here
4. Patients must have organ and marrow function meeting the criteria below:

   Absolute neutrophil count > 2,000/mcL Hemoglobin > 9.0 mg/mL Platelets > 100,000/mcL Total bilirubin within normal limits or known to be elevated due to a benign conjugation defect such as Gilbert's syndrome, as evidenced by normal conjugated bilirubin level AST/ALT < 3X institutional normal limits Creatinine clearance (CrCl) > 50 mL/min/1.73m2, as measured with 24 hr urine collection or estimated by CKD-EPI, whichever is greater
5. Signed, written informed consents to allow transfer of tumor tissue and production of peptides and to receive experimental treatment and monitoring if agreeable, or monitoring without experimental treatment otherwise
6. Age ≥18 years
7. Available fresh tissue from surgical excision. If fresh tissue is not available, archival tissue may be used.
8. Female subjects of childbearing potential must have a negative serum pregnancy test at screening (within 72 hours of first dose of study medication). Non-childbearing potential (other than by medical reasons) is defined as 1 of the following:

   1. ≥ 45 years of age and amenorrheic for >1 year by self-report.
   2. Amenorrheic for >2 years without a hysterectomy and oophorectomy, and follicle-stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation.
   3. Status post-hysterectomy, -oophorectomy, or -tubal ligation. If of childbearing potential, female subjects must be willing to use adequate birth control during the study, starting with the screening visit through 120 days after the last dose of study therapy.

Male subjects with a female partner(s) of childbearing potential must agree to use a condom throughout the trial, starting with the screening visit through 120 days after the last dose of study therapy. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

Note: Abstinence is acceptable for both female and male subjects if this is the subject's established and preferred contraception method.

Exclusion Criteria

1. Subjects must not have previously received a checkpoint inhibitor ie, anti-PD-1, anti-PD L1, or anti CTLA-4 antibody.
2. Subjects must not have previously received anticancer medications or investigational drugs for the disease under study within the following windows:

   a. ≤ 28 days for prior monoclonal antibody used for anticancer therapy, with the exception of denosumab b. ≤ 7 days for immunosuppressive treatment for any reason, with the following exceptions: i. Physiologic steroid replacement for adrenal insufficiency (e.g., <10 mg prednisone per day) is permitted.

   ii. Use of inhaled or topical corticosteroid for radiographic procedures is permitted.

   c. Systemic corticosteroids < 7 days are not allowed except as defined above. d. ≤ 28 days before first dose of study drug for all other investigational study drugs or devices
3. Has persisting toxicity related to prior therapy of National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE) Grade >1 severity.

   Note: Sensory neuropathy or alopecia of Grade ≤2 is acceptable.
4. Has known severe hypersensitivity reactions to fully human monoclonal antibodies (NCI-CTCAE Version 5.0 Grade ≥3), any history of anaphylaxis, or uncontrolled asthma.
5. Active or history of any autoimmune disease (subjects with diabetes type 1, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible). Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study.
6. Any condition requiring systemic treatment with corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroids doses >10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
7. Uncontrolled intercurrent illness, including but not limited to uncontrolled infection, interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or social situations that would limit compliance with study requirements in the opinion of the treating investigator or medical monitor.
8. History of intolerance or allergic reactions attributed to compounds of similar chemical or biologic composition to AGEN1884 or AGEN2034.
9. Women who are pregnant or breastfeeding.
10. Receipt of a live vaccine within 30 days prior to the first dose of study drug.
11. Inability to adhere to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chethan Ramamurthy, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Mays Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The safety run-in phase will enroll initial subjects who will begin treatment with cisplatin and gemcitabine plus AGEN2034 and AGEN 19884. Dose limiting toxicities will be assessed before beginning Phase ll, Stage 1. Evaluation will occur after 2 cycles of therapy prior to administration of third and fourth cycle therapy and progression to planned surgery. If criteria are met to continue to Stage 2, additional subjects will be enrolled to reach the anticipated total of 36 subjects.
Groups:
- Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies: Patients will be treated and endpoints evaluated:
  AGEN1884: A fully human monoclonal Anti-PD-1 Antibody AGEN2034: A fully human monoclonal Anti-PD-1 Antibody Cisplatin: Alkylating antineoplastic agent Gemcitabine: Antimetabolite antineoplastic agent
Period: Safety Run in Phase
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Started | 4
Completed | 2
Not Completed | 2
Not completed — Progression of disease | 2
Period: Phase II, Stage 1
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Started (No participants were enrolled in the Phase II, Stage I of the study due to early termination of the study) | 0
Completed | 0
Not Completed | 0
Period: Phase ll, Stage 2
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies: Participants enrolled with muscle-invasive bladder cancer.
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 59.75 [43 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Tumor Downstaging of >T2 to pT0
Description: pT0 or pCR (defined as no residual tumor in bladder and lymph nodes on resected specimen). Surgery should be performed within 6 weeks after completing up to 4 cycles (last dose) of neoadjuvant therapy, but can be done up to 10 weeks after treatment ends to be evaluable. Otherwise this patient must be replaced for response evaluation.
Time Frame: Completion of four 21 day cycles (approximately 10 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies: Treatment with the following drugs:
  AGEN1884: A fully human monoclonal Anti-PD-1 Antibody
  AGEN2034: A fully human monoclonal Anti-PD-1 Antibody
  Cisplatin: Alkylating antineoplastic agent
  Gemcitabine: Antimetabolite antineoplastic agent
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Number analyzed (Participants) | 4
Participants | 2

2. Secondary Outcome: Evaluation of Safety and Tolerability of AGEN1884 Plus AGEN2034 Plus Cisplatin and Gemcitabine
Description: Evaluation of safety and tolerability of using Agen1884 plus AGEN2034 plus cisplating and gemcitabine chemotherapy in the neoadjuvant treatment of muscle-invasive bladder cancer prior to radial cystectomy. Number of adverse events assessed between 3-5 using the National Cancer Institution Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0)
Time Frame: Baseline to 90 days
Measure: Number; unit: adverse events
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Number analyzed (Participants) | 4
adverse events | 5

3. Secondary Outcome: Pathologic Downstaging to <T2 Rate
Description: Number of subjects who achieved downstaging of the tumor at completion of the possible 4 chemotherapy cycles.
Time Frame: Baseline to Completion of four 21 day cycles (approximately 10 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Number analyzed (Participants) | 4
Participants | 3

4. Secondary Outcome: Completion of Surgery
Description: Number of subjects that progressed from therapy to surgery
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Number analyzed (Participants) | 4
Participants | 4

5. Secondary Outcome: Progression-free Survival at 1 Year
Description: Number of subjects that survived to 1 year from study start without disease progression
Time Frame: 1 year
Population: Due to early termination of the study, data were not collected for this outcome measure
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Correlate Immune Outcomes
Description: To correlate clinical outcomes with immune and biologic endpoints and identify patient and tumor characteristics that can predict treatment responses
Time Frame: 2 years
Population: Due to early termination, not data were collected for this outcome
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to approximately 5 days after last treatment (approximately 10 weeks)
Arm/Group | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin, Gemcitabine Plus Human Monoclonal Antibodies (N=4)
Anorexia (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increase (Hepatobiliary disorders) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Fatigue (General disorders) | 3 (7)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
Headache (General disorders) | 1 (2)
Hyperkalemia (Renal and urinary disorders) | 1 (1)
Hypertension (General disorders) | 1 (3)
Hypokalemia (Renal and urinary disorders) | 1 (3)
Hypotension (General disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (4)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (5)
Non-cardiac chest pain (General disorders) | 1 (1)
Other (General disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (General disorders) | 1 (1)
White blood cells decreased (Blood and lymphatic system disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT04430036/Prot_SAP_000.pdf